CLINICAL TRIAL: NCT01327339
Title: An Open-label, Multi-centre, Observational, Post-marketing Surveillance to Monitor the Safety of REQUIP(Ropinirole) Administered in Korean Restless Leg Syndrome Patients According to the Prescribing Information
Brief Title: REQUIP RLS Post Marketing Surveillance
Acronym: REQUIP RLS PMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 106207
Record Dates: First submitted 2011-03-03; First posted 2011-04-01 (Estimated); Results first posted 2011-04-01 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ropinirole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects eligible for REQUIP prescription: Male and female subjects who were considered appropriate to be prescribed REQUIP according to the prescribing information will be included in this study.
  Interventions: Drug: Ropinirole

INTERVENTIONS:
Drug: Ropinirole — Basically there is no treatment allocation. Subjects who would be administered of ropinirole at their physician's direction will be enrolled. Dosage regimen will be recommended according to the prescribing information. Subjects will be enrolled consecutively.

SUMMARY:
post-marketing surveillance to monitor safety and efficacy of ropinirole during using of treatment for RLS

DETAILED DESCRIPTION:
This study is a post-marketing surveillance to monitor safety and efficacy of ropinirole during using of treatment for RLS(restless leg syndrome) and identify SAEs, adverse drug reactions, and unexpected AEs not described as precautions or warnings and to identify prognostic factors that have an effect on the AEs and to assess effectiveness of ropinirole in real clinical practices after marketing. The subjects are patients prescribed for ropinirole by the investigators at the sites based on prescription information in normal clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with RLS by the investigator
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol

  * To be contactable over the phone
  * To follow the administration regimen.
* A male or female aged 18 years and more at the time of the first prescription.
* Subjects with no experience of RLS treatment using ropinirole

Exclusion Criteria:

Considering the nature of this non-interventional PMS study, there is no strict exclusion criteria set up. GSK Korea encourage the doctors participating this study to enrol the subjects prescribed with Ropinirole following the locally approved Prescribing Information (Appendix ) The following criteria should be checked at the time of study entry.

* Subjects with hypersensitivity to ropinirole and any excipients
* Female who is during the period of the pregnancy or who are lactating

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects are patients prescribed for ropinirole by the investigators at the sites based on prescription information in normal clinical practices.
Sampling Method: Probability Sample
Enrollment: 755 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Ji-Yun Kim BA, Shin-Young Oh MS, Han-Kyu Lee MD, MS and Dr. Yil-Seob Lee MD, PhD. A Post-marketing Surveillance to Monitor the Safety of Ropinirole (Requip) in Korean Patients with Restless Legs Syndrome. [JPERM]. 2012;5:25-30.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this post-marketing surveillance (PMS) study was to monitor the safety and efficacy of Requip under the real clinical setting after launch.
Groups:
- Requip 0.25 mg, 1 mg, 2 mg: Requip tablet containing ropinirole hydrochloride equivalent to 0.25 milligrams (mg), 1 mg, 2 mg of ropinirole administered once daily. All subjects will be administered of Requip in normal prescription use. Dosage regimen can be changed by the investigator according to the prescribing information.
Period: Overall Study
Arm/Group | Requip 0.25 mg, 1 mg, 2 mg
Started | 755
Completed | 747
Not Completed | 8
Not completed — Protocol Violation | 8

BASELINE CHARACTERISTICS:
Groups:
- Requip 0.25 mg, 1 mg, 2 mg: Requip tablet containing ropinirole hydrochloride equivalent to 0.25 mg, 1 mg, 2 mg of ropinirole administered once daily
Arm/Group | Requip 0.25 mg, 1 mg, 2 mg
Number analyzed (Participants) | 747
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who had been administered the investigational drug at least once and had completed safety assessments.
  Years | 60.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected in members of the ITT Population, comprised of all participants who had been administered the investigational drug at least once and had completed safety assessments.
  Participants
    Female | 440
    Male | 307
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected in members of the ITT Population, comprised of all participants who had been administered the investigational drug at least once and had completed safety assessments.
  participants
    Korean | 747
    Not Korean | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event
Description: An adverse event is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: one month
Population: Intent-to-Treat (ITT) Population: all participants who had been administered the investigational drug at least once and had completed all safety assessments.
Measure: Number; unit: participants
Arm/Group | Requip 0.25 mg, 1 mg, 2 mg
Number analyzed (Participants) | 747
participants | 44
Statistical Analysis 1: Comparison: Requip 0.25 mg, 1 mg, 2 mg; Test type: Superiority or Other; percentage of participants = 5.9, 95% CI 2-sided [4.3 to 7.8] — The estimated value represents the percentage of participants with an adverse event

2. Secondary Outcome: Number of Participants With Any Serious Adverse Event
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening , requires hospitalization or results in prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. For a list of all serious adverse events occurring during the course of the study, see the table entitled "Serious Adverse Events" in the Adverse Event section of the results record.
Time Frame: one month
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Requip 0.25 mg, 1 mg, 2 mg
Number analyzed (Participants) | 747
participants | 3

3. Secondary Outcome: Number of Participants With the Indicated Unexpected Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unexpected adverse events include those not listed in the approved product information and not described as precautions or warnings.
Time Frame: one month
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Requip 0.25 mg, 1 mg, 2 mg
Number analyzed (Participants) | 747
participants
  Weight Decrease | 2
  Thirsty | 1
  Eye Pain | 1
  Saliva Increased | 1
  Melena | 1
  Amnesia | 1
  Appendicitis | 1

ADVERSE EVENTS:
Description: Adverse events were coded by using World Health Organization Adverse Reactions Terminology (WHOART, preferred term level) according to the local regulation.
Arm/Group | Requip 0.25 mg, 1 mg, 2 mg
Serious Adverse Events (participants affected / at risk) | 3/747
Other Adverse Events (participants affected / at risk) | 44/747
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Requip 0.25 mg, 1 mg, 2 mg (N=747)
Melena (Gastrointestinal disorders) | 1
Appendicitis (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Requip 0.25 mg, 1 mg, 2 mg (N=747)
Insomnia (Psychiatric disorders) | 13
Nausea (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Chest Pain (General disorders) | 3
Somnolence (Psychiatric disorders) | 3
Dysesthesia (Nervous system disorders) | 3
Headache (General disorders) | 3
Weight Decrease (Metabolism and nutrition disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Sleep Disturbed (Psychiatric disorders) | 2
Thirsty (Metabolism and nutrition disorders) | 1
Eye Pain (Eye disorders) | 1
Hypotension (Cardiac disorders) | 1
Saliva Increased (Gastrointestinal disorders) | 1
Dystonia (General disorders) | 1
Edema (General disorders) | 1
Tremor, Pain (General disorders) | 1
Amnesia (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.